CLINICAL TRIAL: NCT04423458
Title: The Evaluation of Advanced Ultrasonography Applications in the Assessment of Transplanted Kidney Complications
Brief Title: Evaluation of Advanced US Tools in Assessing Allograft Complications
Status: Completed | Type: Observational
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Other Study IDs: 848 -20HH6053
Record Dates: First submitted 2020-06-05; First posted 2020-06-09 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Renal Failure; Chronic Kidney Diseases; Failure,Kidney; Renal Artery Stenosis; Fibrosis; Complications
Keywords: 3D Ultrasound; US elastography; US MFI; Ultrasound; MRI; CT
MeSH Terms: conditions — Renal Insufficiency; Renal Insufficiency, Chronic; Renal Artery Obstruction; Fibrosis | interventions — Imaging, Three-Dimensional

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Transplanted kidney: No intervention is required. Routine Doppler assessment + 3D scan + Shear wave elastography + MicrFlow Imaging will be immediately recorded afterwards
  Interventions: Device: 3D imaging

INTERVENTIONS:
Device: 3D imaging — The study will focus on the accuracy of ultrasound technology in assessing renal transplants.
  The entire assessment should not take more than 25 minutes.

SUMMARY:
This study evaluates the role of advanced US technology in assessing renal transplants as screening tools such as 3D Ultrasound, Ultrasound SWE, and MFI besides current ultrasound conventional metheds.

DETAILED DESCRIPTION:
This study will focus on monitoring renal after transplantation using all US advanced technology.

Aim one will concentrate on the 3D US in assessing artery stenosis (TRAS) compared to the gold standard.

Aim two focuses on will concentrate on Ultrasound elastography in assessing renal stiffness.

Aim three will compare US colour modes such as PD, CD and MFI to assess renal perfusion in three groups.

Duration: 18 Months; participants will have a patient information sheet; once they are happy to participate, consent will be obtained.

Study data will be entered into a database encrypted and stored in the department. Only the study principal investigator (PI) will know the study database password.

ELIGIBILITY:
INCLUSION CRITERIA

* Patients ≥ 18 years.
* Tx patients.
* Gender.

EXCLUSION CRITERIA

* Prisoners.
* Patients < 18 years.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients having /had kindey transplant
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Peak systolic velocity (cm/s). | 12 weeks
  Pean of the blood flow velocities in the artery/ vein peak systolic velocity ≥200 cm/s velocity difference between pre- and post-stenotic segments of 2:1
Peak systolic velocity ratio (PSVR). | 12 weeks
  High velocity flow at the stenosis site divided by a reference velocity (normal before stenosis)
Resistive Index (RI). | 12 weeks
  An RI less than 0.7 to 0.8 is considered normal, more than that it is indicator of transplant dysfunction.

SECONDARY OUTCOMES:
Volumetric stenosis. | 12 weeks
  Plaque volume is calculated automatically with the aid of software with a package of 3D laptop.
3D GSM. | 12 weeks
  Plaque volume is calculated automatically with the aid of software with a package of 3D laptop.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Aslam, PhD, Study Director — Academic Supervisor
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No